CLINICAL TRIAL: NCT02420184
Title: Treatment of Obstructive Sleep Apnea in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Patrick Hanly, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB15-0055
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Sleep Apnea, Obstructive; Renal Insufficiency, Chronic
MeSH Terms: conditions — Sleep Apnea, Obstructive; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP Therapy (Experimental): Participants will receive standard medical care for CKD as well as CPAP therapy for the duration of the study (1 year).
  Interventions: Device: CPAP
- No CPAP (Placebo Comparator): Participants will receive standard medical care for CKD.
  Interventions: Other: No CPAP

INTERVENTIONS:
Device: CPAP — Participants randomized into the experimental CPAP therapy arm will receive CPAP in addition to their standard medical therapy for CKD. CPAP will be worn whenever the participant sleeps for the duration of the study.
  Other Names: Respironics REMstar AutoA-Flex
  Arms: CPAP Therapy
Other: No CPAP — Participants randomized into the placebo comparator no CPAP arm will receive standard medical therapy for CKD.
  Arms: No CPAP

SUMMARY:
This study is being conducted to determine whether treatment of obstructive sleep apnea (OSA) in patients with chronic kidney disease (CKD) improves kidney function. Half of the participants will receive continuous positive airway pressure (CPAP) treatment for their OSA in addition to their regular CKD treatment, while the other half will only receive their regular CKD treatment.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) and associated hypoxemia during sleep have been associated with a decline in kidney function. The abnormalities in kidney function associated with OSA have been improved by treatment of OSA with continuous positive airway pressure (CPAP), which is a common and effective therapy for OSA. Up to now, clinical research on the impact of OSA on kidney function has been performed on patients without CKD. This study will examine the impact of CPAP therapy on kidney function in patients with CKD.

CKD patients with OSA and nocturnal hypoxemia will be randomized into one of two groups where half will receive treatment of their OSA with CPAP and the other half will not. All participants will have kidney function monitored every 3 months for a year by measurement of serum creatinine and proteinuria. The change in estimated glomerular filtration rate (eGFR) and proteinuria between the two groups will be assessed to determine whether treatment of OSA improves kidney function in patients with CKD.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 3 or 4
* OSA (RDI>5) and nocturnal hypoxemia (SaO2 <90% for >12% of night)

Exclusion Criteria:

* Failure to meet inclusion criteria
* Current therapy with CPAP or supplemental oxygen
* Severe daytime sleepiness reflected by an Epworth Sleepiness Score >15
* Any driver who holds a commercial drivers' license or who reports a recent history (past 6 months) of a road traffic accident
* Severe nocturnal hypoxemia reflected by mean SaO2 <80% during level 3 sleep testing
* Daytime hypoxemia reflected by partial pressure of oxygen in arterial blood (PaO2) less than 60 millimetres of mercury (mmHg) during wakefulness
* Hypoventilation reflected by partial pressure of carbon dioxide in arterial blood (PaCO2) greater than 45 millimetres of mercury (mmHg) during wakefulness
* Central sleep apnea that accounts for >50% of the estimated RDI
* Unable to provide informed consent

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-06; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
eGFR (estimated glomerular filtration rate) | 12 months
  Change in eGFR in CPAP group compared to control group.

SECONDARY OUTCOMES:
ACR (albumin/creatinine ratio) | 12 months
  Change in albumin/creatinine ratio (ACR) in CPAP group compared to control group.
Pittsburgh Sleep Quality Index (PSQI) | 12 months
  The PSQI is a validated, self-reported questionnaire that measures subjective sleep quality by asking patients about difficulties initiating and maintaining sleep. The change in PSQI in CPAP group will be compared to control.
Epworth Sleepiness Scale (ESS) | 12 months
  The ESS is a self-reported questionnaire that measures subjective sleepiness. Patients are asked to rate the tendency to fall asleep in eight passive situations. The change in ESS in the CPAP group will be compared to control
Kidney Disease Quality of Life questionnaire (KDQoL) | 12 months
  The KDQoL focuses on the health concerns of patients with chronic kidney disease26. This has been modified slightly, by omitting 2 questions that ask about dialysis, to make it suitable for the non-dialysis CKD population. The change in KDQoL in the CPAP group will be compared to control.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Hanly, MD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rimke AN, Ahmed SB, Turin TC, Pendharkar SR, Raneri JK, Lynch EJ, Hanly PJ. Effect of CPAP Therapy on Kidney Function in Patients With Chronic Kidney Disease: A Pilot Randomized Controlled Trial. Chest. 2021 May;159(5):2008-2019. doi: 10.1016/j.chest.2020.11.052. Epub 2020 Dec 13. PMID 33316238
- [Derived] Rimke AN, Ahmed SB, Turin TC, Pendharkar SR, Raneri JK, Lynch EJ, Hanly PJ. Effect of CPAP therapy on kidney function in patients with obstructive sleep apnoea and chronic kidney disease: a protocol for a randomised controlled clinical trial. BMJ Open. 2019 Mar 23;9(3):e024632. doi: 10.1136/bmjopen-2018-024632. PMID 30904853